CLINICAL TRIAL: NCT04015154
Title: A Post-Market Clinical Evaluation of the Treatment of Femur Fractures With the Femoral Nail Piriformis Fossa (PF) of the T2 Alpha Femur Antegrade GT/PF Nailing System
Brief Title: A Post-Market Clinical Evaluation of the Treatment of Femur Fractures With the Femoral Nail PF
Status: Active, not recruiting | Type: Observational
Sponsor: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Other Study IDs: T2 Alpha Femur Antegrade PF
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Femoral Fracture
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- T2 Alpha Femoral Nail PF: Subjects in the clinical investigation will undergo placement of the Femoral Nail PF of the T2 Alpha Femur Antegrade GT/PF Nailing System which allows for insertion through the piriformis fossa, according to the Instructions for Use and Operative Technique Manual
  Interventions: Device: Femoral Nail PF of the T2 Alpha Femur Antegrade GT/PF Nailing System

INTERVENTIONS:
Device: Femoral Nail PF of the T2 Alpha Femur Antegrade GT/PF Nailing System — The T2 Alpha Femur Antegrade GT / PF Nailing System is intended for temporary stabilization of bone segments or fragments until bone consolidation has been achieved.

SUMMARY:
This investigation is a prospective, multicenter clinical investigation. It is anticipated that a total of 50 subjects will be enrolled at up to 5 sites. Enrollment is estimated to commence in Q4 of 2018. Neither subjects nor investigators are blinded to treatment and the clinical investigation includes a historical control which will be compared to the Femoral Nail PF of the T2 Alpha Femur Antegrade GT/PF Nailing System.

Total duration of enrollment, 12 month follow-up and analysis is expected to take 29 months. The clinical investigation has been designed to follow the surgeon's standard of care for femur fractured subjects, in addition to a 12 month follow-up visit.

The primary endpoint of this clinical investigation is to confirm efficacy/performance at 12 months, as measured by the Lower Extremity Measure (LEM). Confirmation of efficacy/performance at 12 months will be based on an equal or greater (non-inferior) LEM score result of the Femoral Nail PF of the T2 Alpha Femur Antegrade GT/PF Nailing System compared to the T2 Femur benchmark literature.

DETAILED DESCRIPTION:
The objective of this clinical investigation is to demonstrate the safety and efficacy/performance of the Femoral Nail PF of the T2 Alpha Femur Antegrade GT/PF Nailing System. Efficacy/performance of the procedure will be measured by an equal or greater (non-inferior) Lower Extremity Measure (LEM) score result of the Femoral Nail PF of the T2 Alpha Femur Antegrade GT/PF Nailing System compared to the T2 Femur benchmark literature at 12 months.

In addition, demonstration of bone consolidation in correct alignment will be measured by Investigator assessment by 12 months. Safety of the Femoral Nail PF of the T2 Alpha Femur Antegrade GT/PF Nailing System will be demonstrated through reporting of device related intra-operative and post-operative Adverse Events/incidents by 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a male or non-pregnant female age 18 years or older at the time of surgery;
* Subject is willing and able to give written informed consent and comply with the requirements of this Clinical Investigation Plan;
* Subject is intended to be treated with the Femoral Nail PF of the T2 Alpha Femur Antegrade GT/PF Nailing System in accordance with the following legally cleared/ approved Indications for Use:

Indications for Use:

* Fixation of subtrochanteric, intertrochanteric, ipsilateral neck/shaft, comminuted proximal femoral shaft fractures
* Femoral fixation required as a result of pathological disease
* Temporary stabilization of fractures of the femoral shaft ranging from the femoral neck to the supracondylar regions of the femur
* Open and closed femoral fractures
* Pseudoarthrosis and correction osteotomy
* Pathologic fractures, impending pathologic fractures and tumor resections
* Ipsilateral femur fractures
* Fractures proximal to a total knee arthroplasty
* Nonunions and malunions
* Fractures involving osteopenic and osteoporotic bone

Exclusion Criteria:

* Subject is currently enrolled in or plans to enroll in any concurrent drug and/or device clinical investigation that, in the opinion of the Investigator, may confound results;
* Per the Investigator, the subject is in poor general health or undergoing any concurrent disease that would place the subject in excessive risk to surgery (i.e. significant circulatory problems, cardiac disease).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 50 subjects are to be enrolled in this clinical investigation. Subjects participating in this clinical investigation will be recruited from the investigator's standard subject population, where all subjects presenting for treatment of femoral fractures will be evaluated for clinical investigation participation based on the eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Lower Extremity Measure (LEM) | 12 months
  The primary endpoint of this clinical investigation is to confirm efficacy/performance at 12 months, as measured by the Lower Extremity Measure (LEM). Confirmation of efficacy/performance at 12 months will be based on an equal or greater (non-inferior) LEM score result of the Femoral Nail PF of the T2 Alpha Femur Antegrade GT/PF Nailing System compared to the T2 Femur benchmark literature

SECONDARY OUTCOMES:
Safety will be measured by capturing the incidence rate of device-related adverse events | 12 months
  Incidence of device-related adverse events will be monitored by 12 months through data collection and analyses.
Efficacy/Performance will be measured by demonstration of bone consolidation | 12 months
  Bone consolidation will be assessed by 12 months as measured by Investigator assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Gibson, Study Director — Stryker Trauma and Extremities
Locations (4):
- United States (4):
  - St. Cloud Orthopedic Associates, Ltd, Sartell, Minnesota
  - NYU Langone Medical Center, New York, New York
  - UC Health, Cincinnati, Ohio
  - Inova Fairfax Medical Campus, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: No